CLINICAL TRIAL: NCT04296305
Title: Effect of Opioid Infusion Rate on Abuse Liability Potential and Analgesic Efficacy of Intravenous Hydromorphone Among Inpatients With Cancer Pain: A Randomized Crossover Trial
Brief Title: Effect of Opioid Infusion Rate on Abuse Liability Potential of Intravenous Hydromorphone for Cancer Pain
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-0678; NCI-2020-00732 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0678 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and study staff
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (hydromorphone, placebo) (Experimental): TREATMENT PHASE I: Patients receive hydromorphone IV over 2 minutes and placebo IV over 15 minutes.
  TREATMENT PHASE II: Patients receive hydromorphone IV over 15 minutes and placebo IV over 2 minutes.
  Interventions: Drug: Hydromorphone; Drug: Placebo Administration; Other: Questionnaire Administration
- Group B (hydromorphone, placebo) (Experimental): TREATMENT PHASE I: Patients receive hydromorphone IV over 15 minutes and placebo IV over 2 minutes.
  TREATMENT PHASE II: Patients receive hydromorphone IV over 2 minutes and placebo IV over 15 minutes.
  Interventions: Drug: Hydromorphone; Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Hydromorphone — Given IV after
  Other Names: (-)-Hydromorphone; Dihydromorphinone; Hydromorphon
Drug: Placebo Administration — Given IV after
  Other Names: Inactive Drug
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
In cancer inpatient settings, intravenous (IV) opioids are frequently administered in a bolus fashion in order to obtain immediate pain relief. However, data on the abuse liability (AL) potential of IV opioids in cancer patients is limited. No study has investigated the effect of different IV infusion rates on AL potential in patients receiving parenteral opioids for pain control. This phase IV trial will determine the AL potential of a slow IV hydromorphone (SH) bolus administration compared with a fast IV hydromorphone (FH) bolus administration among inpatients with cancer pain. It will also determine the analgesic efficacy and adverse effect profiles of SH versus FH bolus infusions, and explore the relationship between pharmacogenetics and pharmacokinetic (PK) and pharmacodynamic (PD) effects of hydromorphone. This study will eventually help develop evidence-based guidelines regarding the best style of IV opioid administration which will achieve the most optimal pain control while avoiding the undesirable complication of nonmedical opioid use

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the abuse liability potential of slow intravenous (IV) hydromorphone bolus infusion rate with fast IV hydromorphone bolus infusion rate among inpatients with breakthrough cancer pain (from the "DRUG LIKING" scale of the Drug Effects Questionnaire [DEQ] questionnaire).

SECONDARY OBJECTIVES:

I. To compare the abuse liability potentials of slow IV hydromorphone bolus with fast IV hydromorphone bolus among inpatients with breakthrough cancer pain (from the other scales of the DEQ questionnaire).

II. To compare the analgesic efficacy of slow IV hydromorphone bolus with fast IV hydromorphone bolus among inpatients with breakthrough cancer pain.

III. To compare the adverse effects of slow IV hydromorphone bolus with fast IV hydromorphone bolus among inpatients with breakthrough cancer pain.

IV. To explore the abuse liability potential of slow IV hydromorphone bolus with fast IV hydromorphone bolus among the sub group of patients who achieved successful analgesia, defined as at least a two point or 30% reduction in pain intensity score on a 0-10 scale.

V. To obtain exploratory data regarding the relationship between pharmacogenetics and pharmacokinetic (PK) and pharmacodynamic (PD) effects of hydromorphone.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP A:

TREATMENT PHASE I: Patients concurrently receive IV hydromorphone over 2 minutes and IV placebo over 15 minutes.

TREATMENT PHASE II: Patients are then crossed over to concurrently receive IV hydromorphone over 15 minutes and IV placebo over 2 minutes.

GROUP B:

TREATMENT PHASE I: Patients concurrently receive IV hydromorphone over 15 minutes and IV placebo over 2 minutes.

TREATMENT PHASE II: Patients are then crossed over to concurrently receive IV hydromorphone over 2 minutes and IV placebo over 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with diagnosis of cancer
* History of moderate to severe cancer related pain, defined as Numerical Rating Scale (NRS) pain score >= 4/10
* Receiving no or only on as needed doses of opioids
* Normal cognitive status, defined as a normal state of arousal and an absence of obvious clinical findings of confusion, memory deficits or concentration deficits or a Memorial Delirium Assessment Scale (MDAS) score of < 13
* Ability to read and communicate in the English language
* Written informed consent from patient

Exclusion Criteria:

* Contraindications to opioids, or history of opioid allergy
* Inability to secure IV access
* Known history or evidence of nonmedical opioid use (e.g. abuse, misuse, addiction)
* Oxygen saturations < 92% or respiratory rate < 12 breaths/minute on initial assessment
* Resting heart rate > 120 on initial assessment
* Systolic blood pressure > 180 < 90 mmHg or diastolic pressure > 100 < 60 mmHg on initial assessment
* Patients receiving scheduled chronic opioid therapy (defined as the treatment of pain with opioids for >= 7 days)
* Moderate to severe renal insufficiency (defined as glomerular filtration rate [GFR] < 60 ml/min/1.73 m^2)
* Hepatic insufficiency (defined as alanine aminotransferase [ALT] or aspartate aminotransferase [AST] > 3 times the highest normal value, or total bilirubin > 1.5 times the highest normal value)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Abuse liability potential of SH bolus versus FH bolus (from the "DRUG LIKING" scale of the DEQ questionnaire) | From baseline up to 120 minutes post intervention
  This will be measured by: The difference of peak AL scores (maximum score assessed among the measures at 15, 30, 60, and 120 minutes per participant) of the 'drug LIKING' scale in the DEQ-5 questionnaire between the two treatment groups. (For each patient: difference = Max Scale SH+FP - Max Scale FH+SP). If no evidence of carryover effect, a paired t-test will be used. Otherwise a 2-sample t-test will be used only examining differences during the first period of treatment.

SECONDARY OUTCOMES:
Abuse liability potentials of SH bolus versus FH bolus (from the other scales of the DEQ questionnaire) | From baseline up to 120 minutes post intervention
  This will be measured by: The differences of peak AL scores (maximum score assessed among the measures at 15, 30, 60, and 120 minutes per participant) of the FEEL drug effect, HIGH, DISLIKE and MORE items in the DEQ-5 questionnaire between the two treatment groups. (For each patient: difference = Max Scale SH+FP - Max Scale FH+SP). If carryover effect does not exist, a linear mixed effect model will be fitted for the outcome variable to assess if there is any treatment effect, after taking into account of the "sequence" and "period" effect. A random intercept due to patient will also be included.
Analgesic efficacy | From baseline up to 120 minutes post-intervention
  This will be measured by:
  a) The change in NRS pain intensity scores from baseline to the lowest NRS pain score assessed among the measures 12, 30, 60, and 120 minutes post intervention in each treatment group. Wilcoxon rank-sum test will be used.
  1. Frequency of successful analgesia in each treatment group (successful analgesia is defined as at least a two point or 30% reduction in pain intensity score on a 1-10 scale1). The frequency will be estimated along with 95% confidence intervals. Logistic regression model will be applied to assess the effect of demographics and/or clinical measurements on successful analgesia.
  2. The mean time post-intervention until next analgesic dose is reported in each treatment sequence. Wilcoxon rank-sum test will be used.
Adverse effect | From baseline up to 120 minutes post-intervention
  This will be measured by:
  1. The mean change scores (from baseline to the highest score assessed among the measures 12, 30, 60, and 120 minutes post intervention) of the adverse effects assessment scales. Wilcoxon rank-sum test will be used.
  2. of objective adverse effects (respiratory rate < 12 breaths/ minute, O2sat < 94%, SBP< 90mmHg, heart rate > 120 beats per minute) for each treatment group. Frequency and proportion of objective adverse effects will be reported and tabulated. Chi-squared test or Fisher's exact test, whichever appropriate, will be applied to test the association of adverse effect and treatment group.
Abuse liability potential among patients who achieved successful analgesia | From baseline up to 120 minutes post-intervention
  This will be measured by: The peak scores of the five items in the DEQ-5 questionnaire for each treatment group among the subgroup of patients who achieved successful analgesia (defined as at least a two point or 30% reduction in pain intensity score on a 1-10 scale). Wilcoxon rank-sum test will be used.
Plasma concentration (Cmax) and peak (maximal) plasma concentration (Tmax) of hydromorphone metabolite H3G | From baseline up to 120 minutes post-intervention
  This will be measured by estimating the mean Cmax and mean Tmax of hydromorphone and H3G in each treatment group among the measures at 15, 30, 60, and 120 minutes post intervention in each treatment group
Elimination half-life (T1/2) of hydromorphone and its metabolite H3G | From baseline up to 120 minutes post-intervention
  This will be measured by estimating the mean T1/2 of hydromorphone and H3G among the measures at 15, 30, 60, and 120 minutes post intervention in each treatment group
Area-under-the-curve (AUC) of hydromorphone and its metabolite H3G | From baseline up to 120 minutes post-intervention
  This will be measured by estimating the mean AUC of hydromorphone and H3G among the measures at 15, 30, 60, and 120 minutes post intervention in each treatment group
Metabolic ratio of H3G to hydromorphone | From baseline up to 120 minutes post-intervention
  This will be measured by estimating the mean metabolic ratio of H3G to hydromorphone among the measures at 15, 30, 60, and 120 minutes post intervention in each treatment group
Wild-type or single nucleotide polymorphisms (SNiPs) in UGT enzymes in the study population | From baseline up to 120 minutes post-intervention
  This will be measured by calculating number of wild-type or single nucleotide polymorphisms (SNiPs) in UGT enzymes in the study population

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Arthur, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT04296305/ICF_000.pdf